CLINICAL TRIAL: NCT02556814
Title: A Prospective, Multicenter, Placebo Controlled Study on Caffeic Acid Tablet Combining High-dose Dexamethasone in Management of Adult Primary Immune Thrombocytopenia (ITP)
Brief Title: Caffeic Acid Combining High-dose Dexamethasone in Management of ITP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITP-Caffeic acid + HD-DXM
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2018-10

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; Caffeic Acid; dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — caffeic acid; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- caffeic acid tablet and dexamethasone (Experimental): Oral administration of caffeic acid tablets 0.3g three times per day for 3 months. Oral administration of dexamethasone 40 mg for four consecutive days then proceed another cycle 10 days later.
  Interventions: Drug: Caffeic acid tablets; Drug: Dexamethasone
- Placebo and dexamethasone (Active Comparator): Oral administration of placebo tablets 0.3g three times per day for 3 months. Oral administration of dexamethasone 40 mg for four consecutive days then proceed another cycle 10 days later.
  Interventions: Drug: Dexamethasone; Drug: placebo

INTERVENTIONS:
Drug: Caffeic acid tablets — Oral administration of caffeic acid tablets 0.3g three times per day for 3 months
  Other Names: Caffeic acid tablet
  Arms: caffeic acid tablet and dexamethasone
Drug: Dexamethasone — Oral administration of dexamethasone 40 mg for four consecutive days then proceed another cycle 10 days later.
Drug: placebo — Oral administration of placebo tablets 0.3g three times per day for 3 months
  Arms: Placebo and dexamethasone

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of caffeic acid tablets combining with high-dose dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, randomized, double blinded placebo-controlled trial of 240 primary ITP adult patients from 8 medical centers in China. One part of the participants are randomly selected to receive caffeic acid tablets (given orally at a dose of 900mg per day for 3 consecutive months), combining with dexamethasone (given orally at a dose of 40 mg per day for 4 days, two cycles with an interval of 10 days); the others are selected to receive high-dose of dexamethasone treatment plus placebo.

Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of caffeic acid tablets combining with high-dose dexamethasone therapy for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

* 1.Meet the diagnostic criteria for immune thrombocytopenia; 2.Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years; 3.To show a platelet count <30 * 10^9/L, and with bleeding manifestations; 4.Willing and able to sign written informed consent

Exclusion Criteria:

* 1.Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit 2.Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit 3.Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study 4.Current HIV infection or hepatitis B virus or hepatitis C virus infections 5.Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia) 6.Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period 7.Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test 8.Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
sustained response to ITP treatments | 6 months after treatment started
  percentage of patients maintaining PLT count over 30*10^9 without bleeding

SECONDARY OUTCOMES:
Evaluation of platelet response | 3 months after treatment started
  Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD, PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang R, Liu Y, Wang R, Cao J, Hao Y, Xiao T, Yu Z, Yu W, Chu X, Ran X, Zhu C, Xu R, Xiao J, Deng X, Zhang H, Wang Z, Liu G, Hou M, Hou Y. Caffeic acid tablets plus high-dose dexamethasone versus placebo plus high-dose dexamethasone in patients with newly diagnosed immune thrombocytopenia: A multicenter, double-blind, randomized, controlled, phase 2 trial. Chin Med J (Engl). 2025 Aug 22. doi: 10.1097/CM9.0000000000003783. Online ahead of print. PMID 40846660